CLINICAL TRIAL: NCT01915966
Title: Randomized Clinical Trial of a Ginger and Cardamom Gelatin Compared to a Camomile and Lemon Juice Infusion in Control of Xerostomy in Terminally Ill Patients
Brief Title: Efficacy Study of a Ginger and Cardamom Gelatin for Xerostomy in Terminally Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Salut i Envelliment UAB (Other)
Collaborators: Mutuam (Other)
Responsible Party: Principal Investigator, Teresa Peris, Palliativa Care Nurse, Mutuam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FICE-MUT-02-1933-2013
Record Dates: First submitted 2013-07-30; First posted 2013-08-05 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Xerostomia; Salivary Gland Diseases; Mouth Diseases
MeSH Terms: conditions — Xerostomia; Salivary Gland Diseases; Mouth Diseases | interventions — ginger extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardamom, ginger and orange juice gelatin (Experimental): Dietary Supplement
  Interventions: Dietary Supplement: Cardamom, ginger and orange juice gelatin
- Camomile infusion with lemon juice (Active Comparator): Dietary Supplement
  Interventions: Dietary Supplement: Camomile infusion with lemon juice

INTERVENTIONS:
Dietary Supplement: Cardamom, ginger and orange juice gelatin — Patients will receive the recipe of the gelatin, with detailed instructions to prepare it at home, and the necessary ingredients for the gelatin. If necessary, they will be helped in the preparation of an initial batch that should last for one week of treatment. Patients will be instructed to consume the gelatin candy as necessary to alleviate the dry mouth sensation
  Arms: Cardamom, ginger and orange juice gelatin
Dietary Supplement: Camomile infusion with lemon juice — Patients will receive instructions to prepare the infusion at home, and the necessary ingredients. Patients will be instructed to ingest the infusion as necessary to alleviate the dry mouth sensation.
  Arms: Camomile infusion with lemon juice

SUMMARY:
Xerostomia or dry mouth is the subjective feeling that there is not enough saliva in your mouth. It's a frequent symptom in terminally ill patients receiving palliative care, reducing their quality of life and comfort. Usual recommendations in these patients are good oral hygiene and mouthwashes, ad libitum consumption of camomile and lemon juice infusions, and ad libitum sucking of cold (e.g. ice, ice cream) or citric products (e.g. pineapple). Other xerostomia treatments such as artificial saliva and pharmacological drugs (e.g. pilocarpine) are less used in terminally ill patients due to cost and secondary effects.

The purpose of this randomized parallel clinical trial is to determine if a new recipe of gelatin with orange juice, cardamome and ginger is more effective in the control of xerostomia than the usual treatment of camomile infusion with lemon juice against. Treatments will be consumed ad libitum during one week. The main outcome is the subjective assessment of dry mouth at end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Receiving palliative care for terminall illness at MUTUAM PADES
* Complaining of dry mouth and should not have been treated for this problem
* Able to prepare the study supplemental products by himself/herself or having a personal carer willing to do so

Exclusion Criteria:

* Disease of oral mucosa (e.g. oral mycosis, coated oral cavity ).
* Oropharinx neoplasm treated with surgery or radiotherapy.
* Severe cognitive impairment (More than 7 errors in Pfeiffer scale)
* Motor dysphagia causing coordination problems in swallowing.
* Life expectancy less than seven days (Last Days Situation).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Scale of self-perceived mouth dryness (0=not at all, 10=very dry) | At end of treatment (1 week )

SECONDARY OUTCOMES:
Objective signs of xerostomia | At end of treatment (1 week )
  Investigator will assess the presence of xerostomia signs through the assessment of 1) appearance and degree of dryness of tongue, buccal mucosa and lips, and 2)difficulties in speech derived from dry-mouth sensation in the patient.
Scale of subjective assessment of salival disfunction (Pai 2001). | At end of treatment (1 week )
Treatment acceptability | At end of treatment (1 week )
  Participants will answer an open-question regarding their satisfaction with the treatment received, with regards to taste, texture, difficulty of preparation, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Peris, RN, Principal Investigator — Mutuam
Locations (1):
- MUTUAM, Barcelona, Barcelona, Spain